CLINICAL TRIAL: NCT01876433
Title: Beta 3 Agonist Treatment in Heart Failure
Acronym: Beat-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henning Bundgaard (Other)
Responsible Party: Sponsor-Investigator, Henning Bundgaard, Consultant, dr. med., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-004805-29
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction (HFrEF)
MeSH Terms: interventions — mirabegron; Adrenergic beta-3 Receptor Agonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beta-3-agonist (Active Comparator): Mirabegron 25 mg x 2 titrated up to maximal tolerated dosis or a maximum of 150 mg x 2.
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): Placebo 25 mg x 2 titrated up to maximal tolerated dosis or a maximum of 150 mg x 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron
  Other Names: Beta 3 agonist
  Arms: Beta-3-agonist
Drug: Placebo
  Arms: Placebo

SUMMARY:
Objective: The objective of the study is to assess the structural and functional cardiac effects of treatment with the beta 3 AR agonist Mirabegron in patients with chronic heart failure.

Design: The investigators are planning a study aiming at establishing proof of concept that treatment of patients with HF with Mirabegron has significant positive effects, as assessed by clinical and biochemistry measurements, but not by hard endpoints. The investigators are performing a combined dose-finding - chronic efficacy study.

The study is a randomized, placebo-controlled, double-blinded trial. The follow-up period is 6 months. 70 patients with chronic heart failure will be included.

Specific aims

1. Determine safety of administration of Mirabegron to patients with heart failure.
2. Determine if treatment with Mirabegron for 6 months induces beneficial cardiac structural remodelling in patients with heart failure.
3. Determine if Mirabegron improves symptoms and exercise capacity as indicated by questionnaires and 6 min walk test in patients with heart failure.
4. Determine effects of Mirabegron on cardiac conduction, repolarisation and rhythms and arrhythmias in patients with heart failure.
5. Determine effects of Mirabegron on circulating biomarkers in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Stable heart failure NYHA class II-III on ischemic or non-ischemic basis
2. Left ventricular ejection fraction (LVEF) < 40%
3. Stable sinus rhythm (SR)
4. On optimised evidence-based pharmacological HF treatment stable > 4 weeks with no current plan for changing HF therapy. The therapy must include a beta-blocker.
5. No change in diuretics < 4 weeks
6. >18 years

Exclusion Criteria:

1. Unstable cardiac condition
2. Acute myocardial infarction (AMI) or revascularisation < 3 month ago
3. Atrial fibrillation (for technical reasons in relation to imaging and HR reporting)
4. Uncorrected significant primary obstructive valve disease
5. Planned major surgery including cardiac revascularisation
6. Hemodynamically significant obstructive cardiomyopathy
7. Stroke with significant neurological deficit
8. Acute myocarditis or constrictive pericarditis
9. Symptomatic bradycardia or > 1. degree AV-block unless the patient has a pacemaker
10. Clinically significant hepatic (transaminases or bilirubin x 3 above upper reference level) or renal (GFR< 50 ml/min/1,73 m2) diseases
11. Heart failure due to uncorrected thyroid disease
12. Cardiac mechanical support
13. < 6 months after CRT
14. Uncontrolled hypotension (defined as symptomatic systolic blood pressure < 90 mmHg) - or hypertension (defined as systolic at 180 mmHg or above and/or diastolic blood pressure at 110 mmHg or below)
15. Body mass index (BMI) > 35
16. Unable to give informed consent
17. Reduced compliance
18. All women of child bearing potential will be required to use adequate contraception
19. Pregnant or lactating women
20. Treatment with a tricyclic antidepressant or CYP2D6 substrates other than beta-blockers or treatment with digoxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Increase in LVEF (measured by MRI or CT) | 6 months

SECONDARY OUTCOMES:
A reduction in NT proBNP | 6 months
An increase in 6 min walking distance | 6 months
An increase in CO/SV | 6 months
A reduction in LVIDd | 6 months
An improvement in diastolic function | 6 months
A reduction in LA volume | 6 months
A reduction in LV diameters | 6 months
A shortening of the QT interval | 6 months
Improvement in quality of life | 6 monhs
Improvement in functional class | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bundgaard, MD, PhD, DMSc, Principal Investigator — Rigshospitalet Copenhagen University Hospital, Department of Cardiology
Locations (3):
- Australia (2):
  - Monash Center of Cardiovascular Research., Melbourne
  - Department of Cardiology, Royal North Shore Hospital., Sydney
- Department of Cardiology, The Heart Centre, Rigshospitalet Copenhagen University Hospital., Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Bahrami HSZ, Hasselbalch RB, Soholm H, Thomsen JH, Sorgaard M, Kofoed KF, Valeur N, Boesgaard S, Fry NAS, Moller JE, Raja AA, Kober L, Iversen K, Rasmussen H, Bundgaard H. First-In-Man Trial of beta3-Adrenoceptor Agonist Treatment in Chronic Heart Failure: Impact on Diastolic Function. J Cardiovasc Pharmacol. 2024 May 1;83(5):466-473. doi: 10.1097/FJC.0000000000001545. PMID 38452283
- [Derived] Bundgaard H, Axelsson A, Hartvig Thomsen J, Sorgaard M, Kofoed KF, Hasselbalch R, Fry NA, Valeur N, Boesgaard S, Gustafsson F, Kober L, Iversen K, Rasmussen HH. The first-in-man randomized trial of a beta3 adrenoceptor agonist in chronic heart failure: the BEAT-HF trial. Eur J Heart Fail. 2017 Apr;19(4):566-575. doi: 10.1002/ejhf.714. Epub 2016 Dec 18. PMID 27990717